CLINICAL TRIAL: NCT00824291
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study To Evaluate Functional Outcome In Outpatients With Major Depressive Disorder Treated With Desvenlafaxine Succinare Sustained Release
Brief Title: Study Evaluating Desvenlafaxine Succinate Sustained Release In Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3151A1-4415; B2061006
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Results first posted 2010-11-25 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Desvenlafaxine Succinate; Genotype

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: desvenlafaxine succinate sustained release
- 2 (Experimental)
  Interventions: Genetic: Genotyping

INTERVENTIONS:
Drug: desvenlafaxine succinate sustained release — 50 mg/day oral tablet for 12 weeks
  Other Names: Pristiq
  Arms: 1
Genetic: Genotyping — CYP2D6 genotyping at randomization
  Arms: 2

SUMMARY:
This is a multicenter study to assess the health and well-being in subjects who are outpatients with major depressive disorder that take desvenlafaxine succinate sustained release (DVS SR) or placebo for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient men and women, between the ages of 18 to 75 years, fluent in both written and spoken English.
* Employed for 20 hours or more for a minimum of 1 month prior to baseline.
* Primary diagnosis of Major Depressive Disorder with symptoms for at least 30 days prior to baseline.

Exclusion Criteria:

* Treatment with desvenlafaxine succinate sustained release at any time in the past and/or venlafaxine (Effexor or Effexor XR) 1 year prior to baseline.
* Treatment-resistant defined as any of the following failed treatments in the past 3 years: 3 or more previous adequate trials of >=2 classes of antidepressant medication, electroconvulsive therapy, or psychotherapy (2 adequate trials).
* Current (within 12 months prior to the screening visit) psychoactive substance abuse or dependence (including alcohol), manic episode, posttraumatic stress disorder, obsessive-compulsive disorder, or a lifetime diagnosis of bipolar or psychotic disorder.
* Clinically important abnormalities on physical examination, electrocardiogram (ECG), or laboratory evaluations.

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Zilcha-Mano S, Wang X, Wajsbrot DB, Boucher M, Fine SA, Rutherford BR. Trajectories of Function and Symptom Change in Desvenlafaxine Clinical Trials: Toward Personalized Treatment for Depression. J Clin Psychopharmacol. 2021 Sep-Oct 01;41(5):579-584. doi: 10.1097/JCP.0000000000001435. PMID 34183490
- [Derived] Soares CN, Zhang M, Boucher M. Categorical improvement in functional impairment in depressed patients treated with desvenlafaxine. CNS Spectr. 2019 Jun;24(3):322-332. doi: 10.1017/S1092852917000633. Epub 2017 Nov 15. PMID 29140227
- [Derived] Reddy S, Fayyad R, Edgar CJ, Guico-Pabia CJ, Wesnes K. The effect of desvenlafaxine on cognitive functioning in employed outpatients with major depressive disorder: a substudy of a randomized, double-blind, placebo-controlled trial. J Psychopharmacol. 2016 Jun;30(6):559-67. doi: 10.1177/0269881116631649. Epub 2016 Mar 23. PMID 27009044
- [Derived] McIntyre RS, Fayyad R, Mackell JA, Boucher M. Effect of metabolic syndrome and thyroid hormone on efficacy of desvenlafaxine 50 and 100 mg/d in major depressive disorder. Curr Med Res Opin. 2016;32(3):587-99. doi: 10.1185/03007995.2015.1136603. Epub 2016 Jan 13. PMID 26709542
- [Derived] McIntyre RS, Fayyad RS, Guico-Pabia CJ, Boucher M. A Post Hoc Analysis of the Effect of Weight on Efficacy in Depressed Patients Treated With Desvenlafaxine 50 mg/d and 100 mg/d. Prim Care Companion CNS Disord. 2015 Jun 4;17(3):10.4088/PCC.14m01741. doi: 10.4088/PCC.14m01741. eCollection 2015. PMID 26644956
- [Derived] Thase ME, Fayyad R, Cheng RF, Guico-Pabia CJ, Sporn J, Boucher M, Tourian KA. Effects of desvenlafaxine on blood pressure in patients treated for major depressive disorder: a pooled analysis. Curr Med Res Opin. 2015 Apr;31(4):809-20. doi: 10.1185/03007995.2015.1020365. Epub 2015 Mar 26. PMID 25758058
- [Derived] Endicott J, Lam RW, Hsu MA, Fayyad R, Boucher M, Guico-Pabia CJ. Improvements in quality of life with desvenlafaxine 50mg/d vs placebo in employed adults with major depressive disorder. J Affect Disord. 2014 Sep;166:307-14. doi: 10.1016/j.jad.2014.05.011. Epub 2014 May 21. PMID 25012446
- [Derived] Lam RW, Endicott J, Hsu MA, Fayyad R, Guico-Pabia C, Boucher M. Predictors of functional improvement in employed adults with major depressive disorder treated with desvenlafaxine. Int Clin Psychopharmacol. 2014 Sep;29(5):239-51. doi: 10.1097/YIC.0000000000000031. PMID 24583567
- [Derived] Soares CN, Endicott J, Boucher M, Fayyad RS, Guico-Pabia CJ. Predictors of functional response and remission with desvenlafaxine 50 mg/d in patients with major depressive disorder. CNS Spectr. 2014 Dec;19(6):519-27. doi: 10.1017/S1092852914000066. Epub 2014 Feb 26. PMID 24571916
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A1-4415&StudyName=Study%20Evaluating%20Desvenlafaxine%20Succinate%20Sustained%20Release%20In%20Outpatients%20With%20Major%20Depressive%20Disorder

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 752 potential participants were screened for this study. 437 participants were randomized to treatment groups while 315 participants were not randomized (288: did not meet the study criteria; 27 were not randomized for other reasons). Of the 437 randomized participants, 10 participants did not receive the study treatment.
Groups:
- DVS SR 50 mg: Participants were administered an oral dose of Desvenlafaxine Succinate Sustained Release (DVS SR) 50 mg tablet once daily with or without food.
- Placebo: Participants were administered an oral dose of placebo once daily with or without food.
Period: Overall Study
Arm/Group | DVS SR 50 mg | Placebo
Started | 285 | 142
Completed | 231 | 107
Not Completed | 54 | 35
Not completed — Adverse Event | 15 | 6
Not completed — Discontinuation of Study by Sponsor | 1 | 2
Not completed — Lost to Follow-up | 11 | 9
Not completed — Non-compliance | 1 | 1
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 14 | 8
Not completed — Lack of Efficacy | 7 | 8
Not completed — Participant on prohibited medication | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DVS SR 50 mg | Placebo | Total
Number analyzed (Participants) | 285 | 142 | 427
Age Continuous [Mean (Standard Deviation); unit: years] | 43.16 (11.72) | 41.57 (12.64) | 42.63 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 93 | 281
  Male | 97 | 49 | 146

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Depression Scale (HAM-D) at Week 12
Description: HAM-D, clinician-rated interview, measures presence of depressive symptoms in 17 areas (symptoms such as depressed mood, guilt feelings, suicide, sleep disturbances, anxiety levels and weight loss). Total score ranges from 0 to 52; higher scores indicate more depression. Change from baseline: mean at observation minus mean at baseline.
Time Frame: At Baseline and Week 12.
Population: Intent-to-treat (ITT) analysis set, Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DVS SR 50 mg | Placebo
Number analyzed (Participants) | 285 | 142
Scores on a scale | -12.61 (0.45) | -10.50 (0.60)
Statistical Analysis 1: Comparison: DVS SR 50 mg vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Net) = 2.12, 95% CI 2-sided [0.78 to 3.46]

2. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Week 12
Description: Participant rated scale was used to assess the effect of the participant's symptoms on their work/social/family life. Total scores range from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life. Individual item scores range from 0 to 10.
Time Frame: At Baseline and Week 12.
Population: ITT, LOCF
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DVS SR 50 mg | Placebo
Number analyzed (Participants) | 285 | 142
Scores on a scale | -9.41 (0.48) | -8.08 (0.63)
Statistical Analysis 1: Comparison: DVS SR 50 mg vs Placebo; Test type: Superiority or Other; p = 0.067, ANCOVA; Mean Difference (Net) = 1.33, 95% CI 2-sided [-0.09 to 2.76]

3. Secondary Outcome: Clinical Global Impression Scale - Improvement (CGI- I) Score at Week 12
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected. Change = score at observation minus score at baseline.
Time Frame: At Baseline and Week 12.
Population: ITT, LOCF
Measure: Number; unit: Scores on a scale
Arm/Group | DVS SR 50 mg | Placebo
Number analyzed (Participants) | 285 | 142
Scores on a scale
  1 (Very Much Improved) | 103 (0.07) | 31 (0.10)
  2 (Much Improved) | 84 | 44
  3 (Minimally Improved) | 53 | 31
  4 (No Change) | 34 | 30
  5 (Minimally Worse) | 10 | 5
  6 (Much Worse) | 0 | 1
  7 (Very Much Worse) | 1 | 0
Statistical Analysis 1: Comparison: DVS SR 50 mg vs Placebo; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Clinical Global Impressions Scale - Severity of Illness (CGI-S) at Week 12
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected. Change: score at observation minus score at baseline.
Time Frame: At Baseline and Week 12.
Population: ITT, LOCF
Measure: Number; unit: Scores on a scale
Arm/Group | DVS SR 50 mg | Placebo
Number analyzed (Participants) | 285 | 142
Scores on a scale
  1 (Very Much Improved) | 69 (0.08) | 23 (0.11)
  2 (Much Improved) | 68 | 30
  3 (Minimally Improved) | 77 | 31
  4 (No Change) | 56 | 43
  5 (Minimally Worse) | 14 | 15
  6 (Much Worse) | 1 | 0
  7 (Very Much Worse) | 0 | 0
Statistical Analysis 1: Comparison: DVS SR 50 mg vs Placebo; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel

5. Secondary Outcome: Change From Baseline on Work and Activities Item of HAM-D17 at Week 12
Description: The Work and Activities Item of the HAM-D17 is item 7 of HAM-D17. Scoring range from 0 to 4.
Time Frame: At Baseline and Week 12.
Population: ITT, LOCF
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DVS SR 50 mg | Placebo
Number analyzed (Participants) | 285 | 142
Scores on a scale | -1.68 (0.07) | -1.45 (0.10)
Statistical Analysis 1: Comparison: DVS SR 50 mg vs Placebo; Test type: Superiority or Other; p = 0.040, ANCOVA; Mean Difference (Net) = 0.23, 95% CI 2-sided [0.01 to 0.44]

6. Secondary Outcome: Change From Baseline in Adjusted Mean on Montgomery-Asberg Depression Rating Scale (MADRS) at Week 12
Description: Measures the overall severity of depressive symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: At Baseline and Week 12.
Population: ITT, LOCF
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DVS SR 50 mg | Placebo
Number analyzed (Participants) | 265 | 125
Scores on a scale | -18.44 (0.69) | -16.18 (0.94)
Statistical Analysis 1: Comparison: DVS SR 50 mg vs Placebo; Test type: Superiority or Other; p = 0.035, ANCOVA; Mean Difference (Net) = 2.26, 95% CI 2-sided [0.16 to 4.37]

7. Secondary Outcome: Change From Baseline on Worry Anxiety Tension Scale (WATS) at Week 12
Description: WATS: a self-administered, 3-question rating scale assesses worry, anxiety, and tension. Each item was a visual analog scale on which the participant circles a number from 0 to 10. Higher scores indicated worse function. WATS total score was the sum of the 3 items. If 1 item was missing, the total score would be missing.
Time Frame: At Baseline and Week 12.
Population: ITT, LOCF
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DVS SR 50 mg | Placebo
Number analyzed (Participants) | 285 | 142
Scores on a scale | -13.39 (0.79) | -10.95 (1.04)
Statistical Analysis 1: Comparison: DVS SR 50 mg vs Placebo; Test type: Superiority or Other; p = 0.041, ANCOVA; Mean Difference (Net) = 2.44, 95% CI 2-sided [0.10 to 4.78]

8. Secondary Outcome: Change From Baseline on Stress and Social Support Scales at Week 12
Description: Stress and Social Support Scales: self-administered rating scale where item 1 is the stress vulnerability scale measuring how much the subject was set back by stressful events on an 11-point scale ranging from 0 (not at all) to 10 (extremely) and item 2 is an 11-point scale ranging from 0 to 100 percent of the amount of support the subject received from relatives and friends.
Time Frame: At Baseline and Week 12.
Population: ITT, LOCF
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DVS SR 50 mg | Placebo
Number analyzed (Participants) | 285 | 142
Scores on a scale | -2.53 (0.18) | -2.14 (0.23)
Statistical Analysis 1: Comparison: DVS SR 50 mg vs Placebo; Test type: Superiority or Other; p = 0.145, ANCOVA; Mean Difference (Net) = 0.39, 95% CI 2-sided [-0.13 to 0.91]

ADVERSE EVENTS:
Arm/Group | DVS SR 50 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/285 | 2/142
Other Adverse Events (participants affected / at risk) | 213/285 | 90/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR 50 mg (N=285) | Placebo (N=142)
Major depression (Psychiatric disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR 50 mg (N=285) | Placebo (N=142)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 5 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 3 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Blepharospasm (Eye disorders) | 1 | 0
Contact lens intolerance (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 1 | 0
Mydriasis (Eye disorders) | 1 | 0
Photopsia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 2
Visual impairment (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 18 | 11
Diarrhea (Gastrointestinal disorders) | 18 | 10
Dry mouth (Gastrointestinal disorders) | 48 | 9
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Eructation (Gastrointestinal disorders) | 2 | 1
Flatulence (Gastrointestinal disorders) | 3 | 6
Food poisoning (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 56 | 8
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 6 | 4
Asthenia (General disorders) | 3 | 1
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 16 | 5
Feeling abnormal (General disorders) | 0 | 1
Feeling drunk (General disorders) | 0 | 1
Feeling jittery (General disorders) | 5 | 0
Influenza like illness (General disorders) | 1 | 1
Irritability (General disorders) | 3 | 4
Non-cardiac chest pain (General disorders) | 0 | 1
Edema peripheral (General disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 0
Thirst (General disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 1
Bronchitis (Infections and infestations) | 2 | 2
Cystitis (Infections and infestations) | 1 | 1
Ear infection (Infections and infestations) | 2 | 0
Fungal infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 0
Giardiasis (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 3 | 2
Nasopharyngitis (Infections and infestations) | 5 | 3
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 1
Pharyngitis bacterial (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 2
Urinary tract infection (Infections and infestations) | 2 | 2
Vaginal infection (General disorders) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 7 | 4
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 2 | 2
Blood pressure systolic increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Heart rate increased (Investigations) | 1 | 1
Low density lipoprotein increased (Investigations) | 0 | 1
Thyroxine free decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 2
Weight increased (Investigations) | 4 | 4
White blood cell count increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 10 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 3 | 2
Arthralgia (Metabolism and nutrition disorders) | 2 | 2
Back pain (Metabolism and nutrition disorders) | 10 | 2
Bursitis (Metabolism and nutrition disorders) | 1 | 0
Flank pain (Metabolism and nutrition disorders) | 1 | 1
Joint stiffness (Metabolism and nutrition disorders) | 1 | 1
Joint swelling (Metabolism and nutrition disorders) | 2 | 2
Muscle spasms (Metabolism and nutrition disorders) | 4 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Crying (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 28 | 6
Dizziness postural (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 0
Fine motor delay (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 43 | 21
Hypersomnia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 2 | 0
Migraine (Nervous system disorders) | 4 | 2
Paresthesia (Nervous system disorders) | 5 | 1
Presyncope (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 4 | 0
Sinus headache (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 18 | 3
Syncope (Nervous system disorders) | 1 | 1
Tension headache (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 5 | 0
Abnormal dreams (Psychiatric disorders) | 2 | 3
Anorgasmia (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 4 | 1
Bereavement reaction (Psychiatric disorders) | 1 | 0
Bruxism (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0
Initial insomnia (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 13 | 5
Libido decreased (Psychiatric disorders) | 5 | 0
Libido increased (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1
Middle insomnia (Psychiatric disorders) | 2 | 0
Nervousness (Psychiatric disorders) | 1 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0
Violence-related symptom (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Pollakiuria (Psychiatric disorders) | 2 | 1
Breast discharge (Reproductive system and breast disorders) | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 1 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 1
Ejaculation delayed (Reproductive system and breast disorders) | 2 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 4 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 2 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Yawning (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Hot flush (Vascular disorders) | 4 | 2
Hypertension (Vascular disorders) | 9 | 0
Hypotension (Vascular disorders) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tri-iodothyronine decreased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.